CLINICAL TRIAL: NCT01467999
Title: Open-Label Pilot Study of Guanfacine-Extended Release for the Treatment of Cannabis Dependence
Acronym: GUAN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #6393; 6393 (Other: NYSPI IRB)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Cannabis Dependence
Keywords: cannabis dependence; marijuana dependence; guanfacine
MeSH Terms: conditions — Marijuana Abuse | interventions — Guanfacine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Guanfacine (Experimental): Guanfacine, 4mg given once daily
  Interventions: Drug: Guanfacine

INTERVENTIONS:
Drug: Guanfacine — Guanfacine, 4mg given once daily
  Other Names: Intuniv

SUMMARY:
The purpose of this study is to determine whether guanfacine represents a tolerable, potentially effective pharmacotherapy option for cannabis dependence. Interested in seeing whether guanfacine treatment reduces marijuana consumption, withdrawal symptoms, and craving as compared to baseline.

DETAILED DESCRIPTION:
Cannabis use disorders remain the most common illicit drug use disorder and options for treatment remain limited. Compared to other abusable substances, there has been little investigation of pharmacotherapies for cannabis dependence and no effective pharmacotherapy for cannabis dependence has been developed yet. As such, the development of effective cannabis dependence pharmacotherapy is an important unmet public health need. Lofexidine, an alpha-2 agonist, is effective in treating opioid withdrawal and shows promise as cannabis use disorder pharmacotherapy, though its use may be limited by a cumbersome (thrice daily) dosing regimen. An alpha-2-agonist with a longer half-life, such as guanfacine, may have some of the same benefits as lofexidine at comparable doses, but its easier (once daily) dosing regimen may promote compliance and treatment retention. The purpose of this study is therefore to determine whether guanfacine represents a tolerable, potentially effective pharmacotherapy option for cannabis dependence. This pilot study can also provide the basis for subsequently conducting a larger study aimed at determining efficacy with the appropriate randomized, placebo-controlled design.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 18-60 who meet DSM-IV criteria for current marijuana dependence
* Individuals must report using marijuana at least 20 days in the past 30 days and have a positive urine test for THC on the day of study entry.
* Individual must describe marijuana as their primary drug of abuse.
* Individuals must be capable of giving informed consent and capable of complying with study procedures.

Exclusion Criteria:

* Meets DSM-IV-TR criteria for schizophrenia, schizoaffective illness, psychotic disorder other than transient psychosis due to drug abuse, major depression, bipolar illness or psychiatric disorders (other than substance abuse) which require psychiatric intervention.
* Unstable medication conditions, such as poorly controlled diabetes or hypertension (>140/90 mmHg), which might make participation hazardous.
* Individuals with liver enzyme function tests greater than three times normal, or acute hepatitis
* Individuals with a history of a seizure disorder
* Individuals with current suicidal risk.
* Individuals who are cognitively impaired
* Bradycardia (< 50 beats/minute), hypotension (sitting or standing BP < 90/50), or symptoms attributable to low BP (i.e. lightheadedness or dizziness on standing).
* Nursing mothers and pregnant women. Women of child bearing age will be included in the study provided that they are not pregnant, based on the results of a blood pregnancy test drawn at the time of screening. They must also agree to use a method of contraception with proven efficacy and agree not to become pregnant during the study. To confirm this, urine pregnancy tests will be repeated monthly. Women will be provided a full explanation of the potential dangers of pregnancy while on the study medication. If a woman becomes pregnant, the study medication will be discontinued.
* Individuals who are physiologically dependent on any other drugs (excluding nicotine) that would require a medical intervention
* Individuals with known sensitivity to alpha-2 Agonists
* Individuals with coronary vascular disease as indicated by history or suspected by abnormal ECG or history of cardiac symptoms
* Individuals currently being treated with antihypertensive medication, including alpha-2 agonists
* Individuals currently taking medications that may interact adversely with guanfacine.
* Individuals who are court-mandated to treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-02; Primary Completion 2016-04 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances Levin, M.D., Principal Investigator — Columbia University; Elias Dakwar, M.D., Principal Investigator — Columbia University
Locations (1):
- STARS, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants responded to newspapers, radio and public service announcements in the New York City area, and reported at least 20 days of use in the past 30 days.
Period: Overall Study
Arm/Group | Guanfacine
Started | 22
Completed | 9
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Guanfacine
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 5
  More than one race | 6
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Mean Number of Days of Cannabis Use Per Week
Description: The reduction in cannabis consumption quantified by the number of days of cannabis use per week was assessed, as measured by the Time Line followback, reported week 1 compared to week 8.
Time Frame: Daily cannabis use reported during the 8 week trial or the length of the patient's participation
Population: intent-to-treat sample
Measure: Mean (Standard Deviation); unit: days of use per week
Arm/Group | Guanfacine
Number analyzed (Participants) | 22
days of use per week
  week 1 | 4.1 (0.6)
  week 8 | 3.1 (0.9)

ADVERSE EVENTS:
Time Frame: during 8 weeks of open label participation
Arm/Group | Guanfacine
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 14/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guanfacine (N=22)
constipation (Gastrointestinal disorders) | 2 (2)
drowsiness (General disorders) | 3 (3)
dry mouth (General disorders) | 5 (5)
fatigue (General disorders) | 5 (5)
headache (General disorders) | 1 (1)
hypotension (Cardiac disorders) | 3 (3)
increased urination (General disorders) | 1 (1)
insomnia (General disorders) | 5 (5)
lightheadedness (General disorders) | 4 (4)
nausea (Gastrointestinal disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Due to its open-label nature, it is not possible to determine whether the reductions in cannabis use were due to study drug, or whether they were related to other study procedures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No